CLINICAL TRIAL: NCT04722705
Title: Efficacy of Combined Intense Pulsed Light (IPL) With Fractional Erbium:YAG Laser Ablation in Scar Prevention
Brief Title: Combined Intense Pulsed Light (IPL) With Fractional Erbium:YAG Laser Ablation in Scar Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Bo Young Chung, Principal Investigator, Clinical Professor, Hallym University Kangnam Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-11-007
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Intense Pulsed Light; Erbium-yttrium Aluminum Garnet Laser; Scar Prevention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- combined IPL/fractional Er:YAG laser treatment site (Experimental): At baseline, three lesions were randomized to IPL / fractional Er:YAG laser combination therapy site.
  Topical anesthetic cream was applied to the scar 30 minutes before laser treatment. The same dermatologist performed all laser treatments including IPL and 2,940 nm Er:YAG fractional laser. The face was cooled after treatment with gauze soaked in ice water.
  The laser treatment was conducted total three sessions, immediately at suture removal, 4 weeks after suture removal and 8 weeks after suture removal. The evaluation of scar site was conducted 3 months later after last treatment.
  Interventions: Device: fractional Er:YAG laser; Device: Intense pulse light
- fractional Er:YAG laser treatment alone site (Active Comparator): At baseline, three lesions were randomized to fractional Er:YAG laser combination therapy site.
  Topical anesthetic cream was applied to the scar 30 minutes before laser treatment. The same dermatologist performed 2,940 nm Er:YAG fractional laser. The face was cooled after treatment with gauze soaked in ice water.
  The laser treatment was conducted total three sessions, immediately at suture removal, 4 weeks after suture removal and 8 weeks after suture removal. The evaluation of scar site was conducted 3 months later after last treatment.
  Interventions: Device: fractional Er:YAG laser
- untreated control site (No Intervention): At baseline, three lesions were randomized to untreated control site. Topical anesthetic cream was applied to the scar 30 minutes before laser treatment. The evaluation of scar site was conducted 3 months later after last treatment.

INTERVENTIONS:
Device: fractional Er:YAG laser — At baseline, three lesions were randomized. Topical anesthetic cream was applied to the scar 30 minutes before laser treatment.
  The same dermatologist performed 2,940 nm Er:YAG fractional laser. (long pulse mode, 1500mJ, 2Hz, 2 pass) The face was cooled after treatment with gauze soaked in ice water. The laser treatment was conducted total three sessions, immediately at suture removal, 4 weeks after suture removal and 8 weeks after suture removal. The evaluation of scar site was conducted 3 months later after last treatment.
  Other Names: Matrixell, Medro corp., Seoul, Korea
  Arms: combined IPL/fractional Er:YAG laser treatment site; fractional Er:YAG laser treatment alone site
Device: Intense pulse light — At baseline, three lesions were randomized. Topical anesthetic cream was applied to the scar 30 minutes before laser treatment.
  The same dermatologist performed IPL. (irridation energy: 12.5J/cm2, pulse duration: 10ms, 1pass) The face was cooled after treatment with gauze soaked in ice water. The laser treatment was conducted total three sessions, immediately at suture removal, 4 weeks after suture removal and 8 weeks after suture removal. The evaluation of scar site was conducted 3 months later after last treatment.
  Other Names: IPL (Ellipse Flex, DDD, Hoersholm, Denmark)
  Arms: combined IPL/fractional Er:YAG laser treatment site

SUMMARY:
The scar site was divided into 3 sites; combined IPL/fractional Er:YAG laser treatment site, fractional Er:YAG laser treatment site and untreated control site. At baseline, three lesions were randomized to IPL / fractional Er:YAG laser combination therapy site, fractional Er:YAG laser treatment alone site, and untreated control site. The laser treatment was conducted total three sessions, immediately at suture removal (baseline), 4 weeks after suture removal and 8 weeks after suture removal. The evaluation of scar site was conducted 3 months later after last treatment (20 weeks after suture removal).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of postoperative scars on the abdomen
* scars were symmetrical shaped in a line of 3cm or more

Exclusion Criteria:

* uncontrolled systemic or chronic disease
* hypersensitive to the ingredients
* a history of other laser treatments within the past 6 months
* pregnancy
* lactation
* Recent sun exposure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-11-14 (Estimated); Study Completion 2021-11-14 (Estimated)

PRIMARY OUTCOMES:
Patient Observer Scar Assessment Scale | 4 weeks
  The POSAS observer consists of following 6 items: vascularity, pigmentation, thickness, surface area, relief, pliability. Each item was evaluated on a scale from 1 (normal skin) to 10 (worst scar). Finally, the POSAS total score was calculated as the sum of six items, ranging from 6 to 60.
Patient Observer Scar Assessment Scale | 8 weeks
  The POSAS observer consists of following 6 items: vascularity, pigmentation, thickness, surface area, relief, pliability. Each item was evaluated on a scale from 1 (normal skin) to 10 (worst scar). Finally, the POSAS total score was calculated as the sum of six items, ranging from 6 to 60.
Patient Observer Scar Assessment Scale | 20 weeks
  The POSAS observer consists of following 6 items: vascularity, pigmentation, thickness, surface area, relief, pliability. Each item was evaluated on a scale from 1 (normal skin) to 10 (worst scar). Finally, the POSAS total score was calculated as the sum of six items, ranging from 6 to 60.

SECONDARY OUTCOMES:
Total Vancouver Scar scale | 4 weeks
  The VSS consists of 4 following components: vascularity, pigmentation, height ranging from 0 to 3, and pliability from 0 to 5. Score zero means the normal skin, while maximum scores indicate the worst scar.
Total Vancouver Scar scale | 8 weeks
  The VSS consists of 4 following components: vascularity, pigmentation, height ranging from 0 to 3, and pliability from 0 to 5. Score zero means the normal skin, while maximum scores indicate the worst scar.
Total Vancouver Scar scale | 20 weeks
  The VSS consists of 4 following components: vascularity, pigmentation, height ranging from 0 to 3, and pliability from 0 to 5. Score zero means the normal skin, while maximum scores indicate the worst scar.
Erythema index | 4 weeks
  The indexes were measured by placing Spectrophotometer (Cortex Technology, Had- sund, Denmark) directly on the skin lesions for two minutes in the room with constant temperature (20~24 degree Celsius) and humidity (28~38 percent).
  This measurement was performed to determine erythema.
Erythema index | 8 weeks
  The indexes were measured by placing Spectrophotometer (Cortex Technology, Had- sund, Denmark) directly on the skin lesions for two minutes in the room with constant temperature (20~24 degree Celsius) and humidity (28~38 percent).
  This measurement was performed to determine erythema.
Erythema index | 20 weeks
  The indexes were measured by placing Spectrophotometer (Cortex Technology, Had- sund, Denmark) directly on the skin lesions for two minutes in the room with constant temperature (20~24 degree Celsius) and humidity (28~38 percent).
  This measurement was performed to determine erythema.
Melanin index | 4 weeks
  The indexes were measured by placing Spectrophotometer (Cortex Technology, Had- sund, Denmark) directly on the skin lesions for two minutes in the room with constant temperature (20~24 degree Celsius) and humidity (28~38 percent).
  This measurement was performed to determine pigmentation.
Melanin index | 8 weeks
  The indexes were measured by placing Spectrophotometer (Cortex Technology, Had- sund, Denmark) directly on the skin lesions for two minutes in the room with constant temperature (20~24 degree Celsius) and humidity (28~38 percent).
  This measurement was performed to determine pigmentation.
Melanin index | 20 weeks
  The indexes were measured by placing Spectrophotometer (Cortex Technology, Had- sund, Denmark) directly on the skin lesions for two minutes in the room with constant temperature (20~24 degree Celsius) and humidity (28~38 percent).
  This measurement was performed to determine pigmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Young Chung, M.D., PhD, Study Chair — Department of Dermatology, Kangnam Sacred Heart Hospital
Locations (1):
- Kangnam Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No